CLINICAL TRIAL: NCT01616316
Title: Efficacy of Subfascial Approach in Thyroidectomy to Quality of Life in Thyroid Disease Patients: Prospective Randomized Study
Brief Title: Efficacy of Subfascial Approach in Thyroidectomy to Quality of Life in Thyroid Disease Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009-08-058
Record Dates: First submitted 2012-01-18; First posted 2012-06-11 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- subfascial flap (Experimental)
  Interventions: Procedure: subfascial flap
- Subplatysmal flap (Experimental)
  Interventions: Procedure: subplatysmal flap

INTERVENTIONS:
Procedure: subfascial flap — subfacial dissection to thyroid
  Other Names: sub-strap muscle fascial flap approach
  Arms: subfascial flap
Procedure: subplatysmal flap — subplatysmal approach to thyroid
  Other Names: subplatysmal mucle flap approach
  Arms: Subplatysmal flap

SUMMARY:
Subfascial approach method in thyroidectomy maybe result in better quality of life than conventional approach method in thyroid disease patients

ELIGIBILITY:
Inclusion Criteria:

* micropapillary thyroid cancer

Exclusion Criteria:

* lateral neck lymph node metastasis
* severe thyroiditis
* goiter
* reoperation
* extrathyroidal extension

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2010-03; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Dose subfascial approach make better result of swallowing function? | Until 1 year follow up
  To see the effect of subfascial approach for postthyroidectomy swallowing symptom , we will compare the swallowing function between group I(subfascial approach) and group II(subplatysmal approach) after completion of study(after 1 year f/u).
  To check the safety of this study, our result will be checked by korea institutional reveiw board every one year.
Dose subfascial approach make better result of voice symptom? | Until 1 year follow up
  To see the effect of subfascial approach for postthyroidectomy voice function, we will compare the voice function(e.g. hoarseness) between group I(subfascial approach) and group II(subplatysmal approach) after completion of study(after 1 year f/u).
  To check the safety of this study, our result will be checked by korea institutional reveiw board every one year.

SECONDARY OUTCOMES:
The efficacy of subfascial approach in thyroid cancer | Until 1 year follow up
  To see the effect of subfascial approach for postthyroidectomy sensory symptom on neck, we will compare the sensory function and between group I(subfascial approach) and group II(subplatysmal approach) after completion of study(after 1 year f/u).
  To check the safety of this study, our result will be checked by korea institutional reveiw board every one year.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical center, Seoul, South Korea